CLINICAL TRIAL: NCT05685823
Title: The Impact of Conventional Hemodialysis and Renal Transplantation on the Global Longitudinal Strain of the Left Ventricle
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Ureche Carina, MD, Grigore T. Popa University of Medicine and Pharmacy
Other Study IDs: EchoESRD
Record Dates: First submitted 2023-01-08; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Cardiovascular Diseases; Chronic Kidney Diseases; Fibrosis
MeSH Terms: conditions — Cardiovascular Diseases; Renal Insufficiency, Chronic; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to evaluate a group of patients with chronic kidney disease in stages 3-5 by conventional 2D echocardiography, tissue Doppler techniques and speckle tracking - LV GLS and determine the correlation of ultrasound parameters with mortality. Additionally, fibrosis-related biomarkers will be studied in this population.

ELIGIBILITY:
Inclusion Criteria:

* eGFR < 15 ml/min/1.73m2 (CKD - EPI)
* NYHA class I-II
* Hemodynamic stability

Exclusion Criteria:

* age < 18 years old
* poor acoustic window
* atrial fibrillation
* recent Acute Myocardial Infarction
* pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced chronic kidney disease, pre-dialysis or pre-transplant, in the records of the Clinical Hospital "Dr. C. I. Parhon" Iasi
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Variation of GLS | 3 years
All-cause mortality | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Gr T Popa University of Medicine and Pharmacy, Iași, Romania